CLINICAL TRIAL: NCT01829256
Title: Simultaneous Risk Factor Control Using Telehealth to SlOw Progression of Diabetic Kidney Disease (STOP-DKD)
Acronym: STOP-DKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00044811
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Diabetes; Hypertension; Diabetic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacist Telehealth Intervention (Experimental): Will receive a tailored multi-factorial clinical pharmacist-administered telehealth intervention, which includes medication management and behavioral-educational components. The intervention will occur monthly over 3 years.
  Interventions: Behavioral: Pharmacist telehealth intervention
- Education Control (No Intervention): Will receive educational material about management of kidney disease

INTERVENTIONS:
Behavioral: Pharmacist telehealth intervention — A tailored intervention with medication management and behavioral components. The behavioral modules may include, diet, exercise, weight, tobacco use, medication management, side effects, diabetes education, DKD/ HTN/ CVD risk and knowledge.Based on the patient's responses to a series of questions, there will be a provision of tailored feedback to reinforce evidence-based behavior for disease and lifestyle management.
  Arms: Pharmacist Telehealth Intervention

SUMMARY:
Diabetic kidney disease (DKD) is associated with high rates of cardiovascular events and death. In addition, DKD is the major cause of end-stage renal disease (ESRD) in the United States. The purpose of this study is to prevent progression of kidney disease among patients with DKD and uncontrolled hypertension (HTN) using a tailored, telehealth intervention that simultaneously address medication management and modifies multiple risk factors through a combination of patient self-monitoring, behavioral therapies and education to optimize adherence and self-efficacy. Additional goals are to improve control of cardiovascular disease risk factors and reduce cardiovascular events and death.

We hypothesize that patients with DKD and uncontrolled HTN who receive this intervention will have less progression, or a smaller decrease in kidney function, after 3 years when compared to the education control group.

DETAILED DESCRIPTION:
A randomized, controlled trial to slow DKD progression:

1. Using an innovative telehealth approach that is potentially scalable with demonstrable efficacy in reducing antecedents of kidney disease, including poor blood pressure, glucose, and lipid control
2. Enrolling demographically diverse patients from local primary care clinics to allow applicability of our results to the general US population within existing delivery systems; and
3. Targeting patients with moderate DKD (estimated glomerular filtration rate between 45-90 ml/min/1.73m2 with evidence of diabetic nephropathy) and uncontrolled HTN (blood pressure ≥140/90 mm Hg), accounting for about 20% of all patients with diabetes who disproportionately suffer from end-stage renal disease (ESRD), cardiovascular events, and death.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 and less than75 years
* regular use of the Duke University Health System (≥2 primary care visits in 3 prior yrs)
* diagnosis of type 2 diabetes
* have at least 2 serum creatinine values available in the 3 prior years, separated by at least 3 months;
* preserved kidney function (eGFR between 45-90 ml/min/1.73m2 on most recent creatinine)
* evidence of diabetic nephropathy
* uncontrolled HTN (1y mean clinic SBP≥140 and/or DBP≥90).

Exclusion Criteria:

* no access to telephone
* not proficient in English
* nursing home/long-term care facility resident or receiving home health care
* impaired hearing/ speech/ vision
* participating in another trial (pharmaceutical or behavioral)
* planning to leave the area in the next 3 years
* pancreatic insufficiency or diabetes secondary to pancreatitis
* alcohol abuse (>14 alcoholic beverages/ wk)
* diagnosis of non-diabetic kidney disease
* active malignancy (other than non-melanomatous skin cancer)
* life-threatening disease with death probable within 4 years
* Secondary hypertension (renovascular disease, Cushing's syndrome, primary aldosteronism, pheochromocytoma, hypo-/hyperthyroidism, hyperparathyroidism, coarctation of the aorta)
* Pregnancy, Breastfeeding
* Long-term or chronic dialysis
* Dementia
* Renal Transplant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2014-05; Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Change in kidney function as measured by estimated glomerular filtration rate based on cystatin C(eGFRcys) | Measured at Baseline and again at 36 months

SECONDARY OUTCOMES:
Change in blood pressure, glucose/HbA1c and urine albumin | Measured at baseline and again at 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Hayden Bosworth, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System Clinics, Durham, North Carolina, United States

REFERENCES:
- [Derived] Cashmore BA, Cooper TE, Evangelidis NM, Green SC, Lopez-Vargas P, Tunnicliffe DJ. Education programmes for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD007374. doi: 10.1002/14651858.CD007374.pub3. PMID 39171639
- [Derived] Machen L, Davenport CA, Oakes M, Bosworth HB, Patel UD, Diamantidis C. Race, Income, and Medical Care Spending Patterns in High-Risk Primary Care Patients: Results From the STOP-DKD (Simultaneous Risk Factor Control Using Telehealth to Slow Progression of Diabetic Kidney Disease) Study. Kidney Med. 2021 Oct 26;4(1):100382. doi: 10.1016/j.xkme.2021.08.016. eCollection 2022 Jan. PMID 35072046
- [Derived] Zullig LL, Oakes MM, McCant F, Bosworth HB. Lessons learned from two randomized controlled trials: CITIES and STOP-DKD. Contemp Clin Trials Commun. 2020 Jul 8;19:100612. doi: 10.1016/j.conctc.2020.100612. eCollection 2020 Sep. PMID 32685766
- [Derived] Zullig LL, Jazowski SA, Davenport CA, Diamantidis CJ, Oakes MM, Patel S, Moaddeb J, Bosworth HB. Primary Care Providers' Acceptance of Pharmacists' Recommendations to Support Optimal Medication Management for Patients with Diabetic Kidney Disease. J Gen Intern Med. 2020 Jan;35(1):63-69. doi: 10.1007/s11606-019-05403-x. Epub 2019 Oct 28. PMID 31659655
- [Derived] Diamantidis CJ, Bosworth HB, Oakes MM, Davenport CA, Pendergast JF, Patel S, Moaddeb J, Barnhart HX, Merrill PD, Baloch K, Crowley MJ, Patel UD. Simultaneous Risk Factor Control Using Telehealth to slOw Progression of Diabetic Kidney Disease (STOP-DKD) study: Protocol and baseline characteristics of a randomized controlled trial. Contemp Clin Trials. 2018 Jun;69:28-39. doi: 10.1016/j.cct.2018.04.003. Epub 2018 Apr 10. PMID 29649631